CLINICAL TRIAL: NCT02280733
Title: A Longitudinal, Real World, Observational Registry of Chronic Wounds and Ulcers and the Patients Who Have Them
Brief Title: A Real-World Registry of Chronic Wounds and Ulcers
Acronym: WOUNDJOURNEY
Status: Recruiting | Type: Observational
Sponsor: U.S. Wound Registry (Other)
Responsible Party: Sponsor
Other Study IDs: USWR 001
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Foot; Pressure Ulcer; Surgical Wound Dehiscence; Vasculitis; Skin Ulcer; Leg Ulcer; Pyoderma; Peripheral Arterial Disease; Lymphedema; Surgical Complication; Venous Leg Ulcers (VLUs); Calciphylaxis; Sickle Cell Ulcer; Pressure Ulcer (PU); Diabetic Foot Ulcers (DFUs); Pressure Injury; Arterial Ulcers; Soft Tissue Radionecrosis (STRN); Traumatic Wounds; Chronic Ulcer
Keywords: Qualified Clinical Data Registry; Quality Measures; Clinical Data Research Network; Real world data; chronic wounds; chronic ulcers; Diabetic Foot Ulcer; Venous Leg Ulcer; Pressure Ulcer; Pressure Injury; Arterial Ulcer; Traumatic Wound; Surgical Complication; Pyoderma Gangrenosum; Advanced Wound Care; Skin Substitutes; CAMPs; CTPs; Negative Pressure Wound Therapy; NPWT; Collagen Dressings; Compression Therapy; Hyperbaric Oxygen Therapy; Wound Debridement; Real-World Evidence; Comparative Effectiveness; Wound Healing; Amputation; Electronic Health Record (EHR); Debridement; Standard of Care
MeSH Terms: conditions — Diabetic Foot; Pressure Ulcer; Surgical Wound Dehiscence; Vasculitis; Skin Ulcer; Leg Ulcer; Pyoderma; Peripheral Arterial Disease; Lymphedema; Calciphylaxis; Varicose Ulcer; Pyoderma Gangrenosum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- chronic wound patients: This cohort includes pediatric and adult patients with one or more chronic wounds or ulcers treated in any site of care including hospital outpatient clinics, office-based practices, skilled nursing, and home. Data are captured prospectively during routine care using a purpose built certified EHR. Wounds include diabetic foot ulcers, venous leg ulcers, pressure ulcers/injuries, arterial ulcers, surgical wounds, traumatic wounds, and inflammatory ulcers. Interventions are at the discretion of the treating clinician and include standard and advanced wound therapies. Data collected include patient demographics, comorbid conditions, medications, total number of concomitant wounds per patient, wound characteristics, treatments, visit frequency, complications, and outcomes including healing, amputation, recurrence, hospitalization, and death. Patients may be followed for over five years.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Usual care — advanced dressings, off-loading, venous ulcer compression, arterial screening
  Other Names: usual and customary care

SUMMARY:
WOUNDJOURNEY is a longitudinal, real-world, observational registry designed to capture the full clinical course and patient journey associated with chronic wounds and ulcers. Data are collected during routine care from over 1,400 clinicians across the USA and Puerto Rico using a highly structured certified electronic health record (EHR) or electronic data capture (EDC) system. Data are transmitted daily to the U.S. Wound Registry (USWR), a CMS-recognized Qualified Clinical Data Registry (QCDR). The registry captures real-time, research-ready data on patient demographics, comorbidities, wound characteristics, standard-of-care treatments, complications, and advanced therapeutics. It supports robust, fit-for-purpose real-world evidence generation by enabling risk-adjusted outcome analysis, comparative effectiveness research, and quality improvement across diverse sites of care.

DETAILED DESCRIPTION:
WOUNDJOURNEY is a longitudinal, real-world observational registry focused on the chronic disease burden and patient journey of individuals with chronic wounds and ulcers. Data collection began in 2005 and continues prospectively, capturing structured clinical data at the point of care using a purpose-built certified EHR or EDC system. These data are securely transmitted to the U.S. Wound Registry (USWR), a CMS-designated Qualified Clinical Data Registry (QCDR).

All major wound types are represented: Diabetic foot ulcers (DFUs), diabetic ulcers not on the foot, Venous leg ulcers (VLUs), Arterial ulcers, Pressure ulcers/injuries, Surgical complications, Traumatic wounds, Vasculitic/inflammatory, and sickle cell-related ulcers, and chronic non-pressure ulcers.

The registry collects detailed data on standard-of-care practices and advanced wound care interventions, including brand-specific information on: Advanced dressings (e.g., collagen, antimicrobial), Compression therapy, Offloading devices, Cellular and/or tissue-based products (CTPs) also called Cellular, Acellular, or Matrix-like Products (CAMPs) or "skin substitutes," Negative pressure wound therapy, MIST therapy (low-frequency ultrasound), Topical oxygen therapy (TOT), Hyperbaric Oxygen Therapy (HBOT), Topical growth factors (e.g., Becaplermin), Enzymatic and mechanical debridement, Fluorescent imaging for bacterial load, Topical antibiotics and antimicrobials, and other treatments.

The registry captures key elements of the patient journey, including: Frequency of debridement, Sites of care, number of patient visits and number of wound visits, Dressing changes, Use and timing of advanced therapies, Comorbid disease burden and clinical complexity, Patient Frailty, number of wounds and ulcers per patient, patient time in service, wound time service, patient and wound outcomes, the development of new wounds while in service and complication rates.

Wounds are risk stratified using the Wound Healing Index, enabling case-mix adjustment and longitudinal outcome tracking. Follow-up may extend over five years, capturing outcomes such as: Complete healing (epithelialization), Non-healing, Major and minor amputations, Mortality, and Loss to follow-up or transfer of care. Quality of care is assessed using wound-specific quality measures. The registry integrates real-world clinical care with research and quality improvement, supporting a learning healthcare system model.

Through secure tokenization, registry data may be linked to payer claims for comprehensive longitudinal analysis of healthcare utilization, interventions, hospitalizations, medication use, and long-term outcomes across care settings. This enables rigorous, policy-relevant evaluations of standard care and advanced wound therapies in routine practice. The robust patient and wound level data are suitable to understand the natural history of chronic wounds and ulcers and to create historical controls for prospective clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Presence of one or more chronic wounds or ulcers of any etiology
* Wound or ulcer must be treated at a participating site (which can be a hospital outpatient department, office, mobile practitioner, in the home setting, skilled nursing, etc.)
* Care must be documented using the purpose-built, wound-specific structured electronic health record (EHR) or electronic data capture (EDC) system
* All ages, including infants and patients aged 90 years or older (reported in aggregate in accordance with HIPAA de-identification standards)
* All sexes and gender identities
* All wound types and severities, including multiple wounds per patient

Exclusion Criteria:

-None (the registry includes all eligible patients treated at participating sites without sampling or exclusion criteria)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic wounds or ulcers treated at participating sites in any US State and Puerto Rico. All patients and wounds are included without sampling. Each wound can be analyzed independently, even when multiple wounds exist on a single patient.
  Sampling Method:
  Non-Probability Sample
  Minimum Age:
  0 Years
  Maximum Age:
  None (patients aged 90+ are reported in aggregate per HIPAA)
  Sex:
  All
  Gender Based:
  No
  Accepts Healthy Volunteers:
  No
Sampling Method: Non-Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2005-01-01 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Healed | 1 year
  Wound closure by secondary intention
Major amputation | 1 year
  Below the knee, above the knee
Minor amputation | 1 year
  toe amputation, transmetatarsal amputation, midfoot amputation
Patient Death | 1 year
  patient death while in treatment

SECONDARY OUTCOMES:
Percent surface area (PAR) reduction over time | variable - measured at multiple intervals (e.g., 4, 12, 16, 24, and 52 weeks)
  Percent surface area reduction (PSAR) is defined as the percentage decrease in wound surface area from the initial documented size at baseline (first qualifying wound care visit) to subsequent visits over time. Wound surface area is measured using length × width, captured at the point of care using structured fields within the electronic health record (EHR) or electronic data capture (EDC) system. Values are recorded in cm² and used to calculate PSAR as:
  [(Baseline area - Follow-up area) ÷ Baseline area] × 100
  This metric is assessed at multiple time intervals, including 4 weeks, 12 weeks, 16 weeks, 6 months, and 12 months. PSAR is a key performance indicator for healing trajectory and is used to evaluate response to interventions. All wound types are included, and multiple wounds per patient are analyzed independently. Surface area measurements are case-mix adjusted using the Wound Healing Index for comparative effectiveness and quality reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline E Fife, MD, Principal Investigator — Intellicure LLC
Locations (1):
- US Wound Registry, The Woodlands, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) collected through the U.S. Wound Registry (USWR) may be made available to qualified researchers, payers, regulatory agencies, or industry partners upon request. Shared data may include demographics, comorbidities, wound characteristics, interventions, and outcomes captured longitudinally in a structured electronic health record (EHR) or data capture system. All shared data comply with HIPAA de-identification standards and may be subject to data use agreements and institutional review board (IRB) approval.
Time Frame: Available upon request after data quality review and registry updates are complete. IPD is available on an ongoing basis, with no fixed end date.
Access Criteria: Access to de-identified individual participant data (IPD) may be granted to qualified researchers, payers, regulatory agencies, or industry partners upon request. Requests must include a research protocol or data use justification. Data access is contingent on execution of a data use agreement (DUA) and, where applicable, institutional review board (IRB) approval. All shared data will comply with HIPAA de-identification standards (45 CFR §164.514). The U.S. Wound Registry reserves the right to review all requests for scientific merit, relevance, and feasibility. Contact the registry to initiate a data access request. For access inquiries, contact: cfife@intellicure.com

REFERENCES:
- [Background] Fife CE, Walker D, Thomson B, Otto G. The safety of negative pressure wound therapy using vacuum-assisted closure in diabetic foot ulcers treated in the outpatient setting. Int Wound J. 2008 Jun;5 Suppl 2(Suppl 2):17-22. doi: 10.1111/j.1742-481X.2008.00467.x. PMID 18577134
- [Background] Fife CE, Walker D, Thomson B. Electronic Health Records, Registries, and Quality Measures: What? Why? How? Adv Wound Care (New Rochelle). 2013 Dec;2(10):598-604. doi: 10.1089/wound.2013.0476. PMID 24761335
- [Background] Horn SD, Fife CE, Smout RJ, Barrett RS, Thomson B. Development of a wound healing index for patients with chronic wounds. Wound Repair Regen. 2013 Nov-Dec;21(6):823-32. doi: 10.1111/wrr.12107. Epub 2013 Oct 17. PMID 24134202
- [Background] Carter MJ, Fife CE, Walker D, Thomson B. Estimating the applicability of wound care randomized controlled trials to general wound-care populations by estimating the percentage of individuals excluded from a typical wound-care population in such trials. Adv Skin Wound Care. 2009 Jul;22(7):316-24. doi: 10.1097/01.ASW.0000305486.06358.e0. PMID 20375969
- [Background] Fife CE, Carter MJ, Walker D, Thomson B. A retrospective data analysis of antimicrobial dressing usage in 3,084 patients. Ostomy Wound Manage. 2010 Mar 1;56(3):28-42. PMID 20368672
- [Background] Fife CE, Carter MJ, Walker D. Why is it so hard to do the right thing in wound care? Wound Repair Regen. 2010 Mar-Apr;18(2):154-8. doi: 10.1111/j.1524-475X.2010.00571.x. Epub 2010 Feb 16. PMID 20163568
- See also: US Wound Registry Website — http://www.uswoundregistry.com/